CLINICAL TRIAL: NCT06120153
Title: A Cluster-randomized Trial of Point-of-care PCR Diagnostics of Respiratory Tract Infections in General Practice
Brief Title: Point of Care Polymerase Chain Reaction (PCR) Diagnostics of Respiratory Tract Infections in General Practice
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Roche Diagnostics GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: POCPCRdiagnosticsRCT
Record Dates: First submitted 2023-06-26; First posted 2023-11-07 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Respiratory Tract Infections
Keywords: Point of care PCR; General Practice
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Intervention Model Description: Non-blinded cluster randomized cross-over trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- POC PCR-test device (Active Comparator): In the seven-week intervention, the Point-of-Care PCR-testing device will be made available for approximate 50 clinics. Besides the general instructions on how to include patients, clinics in the intervention arm will be instructed that it is entirely up to the GP whether or not to use the PCR-testing device on each individual patient. In addition, no specific instructions on medical treatments or follow up procedures are made.
  Interventions: Diagnostic Test: POC PCR-test device
- Standard testing (No Intervention): In the seven-week control period, the Point-of-Care PCR-testing device will not be available in approximately 50 clinics. Patients attended by the GP during control periods will receive treatment as usual. Like GPs in the intervention arm, GPs in the control arm are not actively encouraged to change their prescription patterns, but they must record data from patients with respiratory tract infections parallel to the intervention group.

INTERVENTIONS:
Diagnostic Test: POC PCR-test device — The analysis will follow an intention-to-treat principle, that is, contacts in the intervention period will be analyzed as randomized, regardless of whether the POC PCR test was actually performed for a given contact. As sensitivity analysis, the data will be analyzed in a "per-protocol" spirit, defining the intervention at the contact level as a POC PCR test performed.
  Arms: POC PCR-test device

SUMMARY:
The present study will assess the effect and cost-effectiveness of the availability of point-of-care (POC) PCR testing, in respiratory tract infections (RTIs) in general practice, compared with usual care.

DETAILED DESCRIPTION:
Background: Respiratory tract infections (RTIs) are frequent reasons for medical consultations and diagnostic accuracy is important to ensure appropriate treatment. It is important for the quality of the healthcare system that patients are diagnosed as fast as possible and that the GP and the patient are reassured about the diagnostic accuracy. If not, the patient may be unnecessarily concerned and contact health services again.

Re-contacts are costly for society, but they may also be unsatisfactory to the patient and the clinician, because many re-contacts may indicate that tentative diagnosis or treatment were not successful and that in some cases the patient needs to contact health services again to get a sufficient answer or to be reassured that nothing is dangerous.

The introduction of POC PCR in primary care settings has demonstrated significant improvements in appropriate antibiotic prescription patterns in high income countries. In Denmark around 88 pct. of all prescription drugs are issued by general practice, as is the vast majority of the total antibiotics consumption in the healthcare system.

Antibiotic overuse may lead to microbial resistance and if the overall consumption is not reduced, infections with resistant bacteria will be a major problem for both patients and healthcare systems. Due to diagnostic uncertainty, GPs may in some situations prescribe antibiotics also in cases where the patient's symptoms are caused by a viral infection.

Further, if antibiotics are not prescribed, the patient may reconsult their GP or the out-of-hours services due to feelings of uncertainty.

Aims: The aim of the study is to evaluate the effect of POC PCR availability in general practice on 1) the number of re-contacts for patients with symptoms of RTIs, 2) the number of hospital admission, 3) deaths, 4) the number of redeemed antibiotic prescriptions, 5) costs, 6) health-related quality-of-life, 7) cost-effectiveness compared to usual care and 8) GP satisfaction.

Furthermore, a qualitative process evaluation will be conducted throughout the trial.

Methods This study is a cluster-randomized crossover, non-blinded superiority trial with a 1:1 allocation ratio. The procedure for randomization takes outset in the clinics' identification numbers as units. The trial consists of two periods of seven weeks (intervention and control). Care-as-usual is used as a comparator. The study is approved by the local regional ethics committee.

The effectiveness study and the cost-effectiveness study will be based on questionnaire data and data from the unique Danish national registries. Information from the different registers will be linked by the patients' Danish Personal Identification Number. Outcomes based on questionnaire data will be collected at baseline, day 7, 14 and day 28 after the initial visit.

GP and patient recruitment:

General practices in 4 out of 5 Danish regions have been invited to participate. GPs have been invited through a written letter and regional newsletters sent to all GPs in Denmark in March 2023. The GPs has been assigned at random to start as intervention or control practice. Based on sample size calculation, the goal was to include 100 GP clinics.

Each practice is asked to register all patients with symptoms of respiratory tract infections consecutively. The GPs are informed that it is entirely up to them and their clinical judgement to make a decision about whether or not they deem it relevant to employ the POC PCR-test device in the consultation with the patient.

ELIGIBILITY:
Inclusion criteria:

* GP clinics are eligible for participation when they have a clinic provider number ("ydernummer").
* Any patient with symptoms of RTI independent of age, gender, socioeconomic factors are eligible for POC PCR testing, if the GP finds it clinically relevant.
* Questionnaire data will be collected from patients ≥15 years old, parents/caregivers to patients ˂15 years and GPs.
* Qualitative data will be collected from consenting patients and/or parents/caregivers to patients <15 years and healthcare staff

Exclusion criteria:

- Questionnaire data of participants below 15 years

Min Age: 0 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 5700 (Estimated)
Dates: Start 2023-10-30 (Actual); Primary Completion 2026-03-22 (Estimated); Study Completion 2026-03-22 (Estimated)

PRIMARY OUTCOMES:
Reduction of respiratory tract infections (RTI) patients' re-contacts to General Practitioners | 2 x 7 weeks of trial = 14 weeks in total (exclusive crossover)
  The primary outcome measure is change in the number of re-contacts within a time period of 7 days from initial contact for each patient consulting with a clinic for a RTI in the intervention period compared to the control period. The re-contacts include any daytime contacts to general practice and are based on data from the national Danish registries. RTI patients may present themselves with symptoms often associated with RTI, e.g., fever, cough, sore throat etc., but it is up to the treating clinician to categorize patients as having a RTI.
  Each time period (i.e., intervention and control) consists of 7 weeks.

SECONDARY OUTCOMES:
Change in number of hospital admission and deaths | Within a time period of 14 days from initial contact for a respiratory tract infection
  Change in number of hospital admission and deaths in the intervention period compared to the control period. Hospital admission and deaths are based on data from the national Danish registries.
Change in number of redeemed antibiotic prescriptions | Within a time period of 7 days from initial contact for a respiratory tract infection
  Change in number of redeemed antibiotic prescriptions in the intervention period compared to the control period. The number of prescriptions are based on data from the national Danish registries.
Effect of POC PCR in general practice on patient satisfaction based on patient satisfaction questionnaires. | On the initial contact for RTI (baseline)
  Effect of POC PCR in general practice on patient satisfaction based on patient satisfaction questionnaires. Satisfaction is measured on a five-point likert scale, ranging from "strongly disagree" to "strongly agree".
Effect of POC PCR in general practice on GP satisfaction based on GP satisfaction questionnaires | At the end of trial (through study completion, an average of 23 weeks)
  Effect of POC PCR in general practice on GP satisfaction based on GP satisfaction questionnaires aimed to be on five point likert scales, but adapted on basis of interviews with participating healthcare personnel. The scales will be ranging from "Strongly disagree" to "Strongly agree".
Total treatment costs 28 days from the initial contact for RTIs based on data from Danish national registers | 28 days from the initial contact for RTI
  The Effect of POC PCR in general practice on healthcare costs based on data from Danish national registers.
Productivity costs based on WPAI-GH-questionnaires | Productivity loss will be measured at baseline (day of the initial visit to the GP for RTI), as well as at day 7, 14 and day 28 after the initial visit.
  The effect of POC PCR in general practice on productivity loss. Measured by (an adjusted version of) Work Productivity and Activity Impairment General Health(WPAI-GH). The WPAI-GH consist of six questions: 1=currently employed; 2=hour missed due to health problems, 3=hours missed other reasons, 4= hours actually worked; 5=degree health affected productivity while working (using a 0 to 10 Visual Analogue Scale (VAS)); 6= degree health affected productivity in regular unpaid activity (0-10 VAS). Answers from the six questions will be combined to estimate the value of productivity loss.
Health-related quality of life (EQ-5D-5L) | HRQoL will be measured at baseline (day of the initial visit to the GP for RTI), as well as at day 7, 14 and day 28 after the initial visit.
  The effect of POC PCR in general practice on Health-related-Quality-of-Life (HRQoL) Health-related-Quality-of-life is assessed with the "EuroQol, 5 Dimensions with 5 Levels" instrument (EQ-5D-5L) with range 5-25 and higher values indicating higher quality of life. The Danish version of the EQ-5D-5L will be used to assess health status in five dimensions (mobility, self-care, daily activities, pain/unease, and anxiety/depression) with five levels of severity (no problems, slight problems, moderate problems, severe problems, and either extreme problems or unable to perform activity).
Cost-effectiveness | Within 28 days
  Cost-effectiveness of POC PCR in general practice Cost effectiveness will be measured according to Incremental cost-effectiveness ratio (ICER).
  Change in cost-effectiveness will be calculated as differences in mean costs divided by the difference in mean number of recontacts.
  For costing, a limited societal perspective will be assumed. Healthcare costs and travel costs will be collected from Danish national registries and productivity loss will assess based on questionnaire data.
Cost-utility | Within 28 days
  Cost-utility of POC PCR in general practice. Cost-utility will be measured according to Incremental cost-effectiveness ratio (ICER).
  Change in cost-utility Cost-utility will be measured by the EuroQol, 5 Dimensions with 5 Levels instrument (EQ-5D-5L) and Danish value sets will be used to calculate Quality-adjusted-life-years (QALYs). QALYs range from 0 to 1, where 0 means dead and 1 means perfect health. The ICER will be calculated as the differences in mean cost divided by the difference in mean QALYs.
  For costing, a limited societal perspective will be assumed. Healthcare costs and travel costs will be collected from Danish national registries and productivity loss will assess based on questionnaire data.
Qualitative process evaluation | Prior and during the 14 weeks study period
  In line with MRC-guidelines, a qualitative assessment and explanation of the factors that could promote or inhibit the uptake of the intervention among health professionals involved in the trial.
  The evaluation focuses on the experience and use of the POC PCR-test in the clinics.
  Methods: 10 pre-intervention interviews with GPs and practice members and 10 post-intervention interviews with GPs and practice members are conducted. Observation studies in 5 clinics before and during trial is conducted. Approximately 15 interviews with patients are conducted.

CONTACTS AND LOCATIONS:
Overall Officials: Jens Søndergaard, MD, PhD, GP, Principal Investigator — University of Southern Denmark
Locations (1):
- Research Unit of General Practice, Dept. of Public Health, University of Southern Denmark, Odense C, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jose BP, Camargos PA, Cruz Filho AA, Correa Rde A. Diagnostic accuracy of respiratory diseases in primary health units. Rev Assoc Med Bras (1992). 2014 Nov-Dec;60(6):599-612. doi: 10.1590/1806-9282.60.06.021. PMID 25650863
- [Background] Vedsted P OF. Almen praksis' funktion og roller. 1 ed. Ehrenreich B MR, Vedsted P, editor. København: Munksgaard; 2011.
- [Background] Cohen JF, Pauchard JY, Hjelm N, Cohen R, Chalumeau M. Efficacy and safety of rapid tests to guide antibiotic prescriptions for sore throat. Cochrane Database Syst Rev. 2020 Jun 4;6(6):CD012431. doi: 10.1002/14651858.CD012431.pub2. PMID 32497279
- [Background] Pottegard A, Olesen M, Christensen B, Christensen MB, Hallas J, Rasmussen L. Who prescribes drugs to patients: A Danish register-based study. Br J Clin Pharmacol. 2021 Jul;87(7):2982-2987. doi: 10.1111/bcp.14691. Epub 2021 Jan 25. PMID 33496033
- [Background] Organization. WH. Global action plan on antimicrobial resistance. Geneva:. World Health Organization; 2015.
- [Background] AI RNM. Improving efficiency in cluster-randomized study design and implementation: taking advantage of a crossover. Open Access Journal of Clinical Trials. 2014;6:11-5.
- [Background] Moore GF, Audrey S, Barker M, Bond L, Bonell C, Hardeman W, Moore L, O'Cathain A, Tinati T, Wight D, Baird J. Process evaluation of complex interventions: Medical Research Council guidance. BMJ. 2015 Mar 19;350:h1258. doi: 10.1136/bmj.h1258. PMID 25791983
- [Background] Foundation. ER. EQ-5D-Y User Guide. 2020.
- [Background] Thygesen LC, Daasnes C, Thaulow I, Bronnum-Hansen H. Introduction to Danish (nationwide) registers on health and social issues: structure, access, legislation, and archiving. Scand J Public Health. 2011 Jul;39(7 Suppl):12-6. doi: 10.1177/1403494811399956. PMID 21898916
- [Derived] Balasubramaniam K, Simonsen LM, Kongstad LP, Thilsing T, Wehberg S, Hallas J, Sopina L, Nielsen JB, Overbeck G, Hvidt EA, Jarbol DE, Rasmussen TL, Sondergaard J. Evaluating the Effect of a Molecular Point-of-Care Test on Acute Respiratory Infections in General Practice: Protocol for a Cluster Randomized Trial. JMIR Res Protoc. 2025 Sep 8;14:e72842. doi: 10.2196/72842. PMID 40921063